CLINICAL TRIAL: NCT03694587
Title: A Single and Multiple Dose, Randomised, Open-label, Cross-over, Healthy Volunteer, Phase I Study of the Pharmacokinetics of a Novel 200 mg Ibuprofen Medicated Plaster
Brief Title: pK of a Novel 200 mg Ibuprofen Medicated Plaster
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medherant Ltd (Industry)
Collaborators: Cooperative Clinical Drug Research and Development AG (CCDRD AG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MED-IBU-101
Record Dates: First submitted 2018-08-16; First posted 2018-10-03 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test IMP (Active Comparator)
  Interventions: Drug: Ibuprofen 200 mg TEPI Medicated Plaster
- Reference IMP (Active Comparator)
  Interventions: Drug: Aktren® 200 mg überzogene Tabletten (Ibuprofen)

INTERVENTIONS:
Drug: Ibuprofen 200 mg TEPI Medicated Plaster — Ibuprofen 200mg TEPI medicated plaster applied to the upper back daily for 24 hours for 5 days
  Arms: Test IMP
Drug: Aktren® 200 mg überzogene Tabletten (Ibuprofen) — one dose of Aktren® 200 mg überzogene Tabletten (Ibuprofen tablet)
  Arms: Reference IMP

SUMMARY:
This is a Phase I study of the pharmacokinetics of a novel 200 mg Ibuprofen Medicated Plaster. The study will be conducted as a monocentric, open, randomised, single and multiple-dose, two-period, crossover trial in healthy volunteers. A total of 16 healthy volunteers will be randomised.

A wash-out period of 3 days is planned between the two periods. Each of the volunteers will be randomly assigned to one of 2 possible administration sequences.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject
* Age between 18 and 65 years
* Physically and mentally healthy as judged by means of medical and standard laboratory examinations
* Non-smokers or ex-smokers (stopped at least 6 months ago) with a smoking history of ≤5 pack-year equivalents (1 pack-year equivalent is equal to smoking 1 pack per day for 1 year**) and non-users of other nicotine containing products, confirmed by urine cotinine test
* Weight ≥ 60 kg and BMI within the range (including the borders)1 of 18.0 to 30.0 kg/m2
* Informed consent given in written form according to chapter 5.4 of the study protocol

Exclusion Criteria:

* Participation in another clinical trial at same time or within the preceding 90 days (calculated from the date of the final examination of the previous study)
* Fertile women without reliable contraception method. List of medically accepted contraceptive methods (used at least 4 weeks prior entry screening visit and not to be changed for the duration of the study):
* combination of 2 barrier methods: female/male condoms, diaphragms, spermicides
* voluntary sterilization (female tubal occlusion).
* Randomisation into the present trial more than once
* Blood donation or blood loss including plasmapheresis of >500 ml in the last 90 days before entry screening
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at entry screening
* History of drug abuse or use of illegal drugs: use of soft drugs, e.g. marihuana within 6 months of entry screening or hard drugs, e.g. cocaine, amphetamines, phencyclidine within 1 year before entry screening
* Alcohol abuse, i.e. regular use of more than 2 units of alcohol per day or 10 units per week or a history of alcoholism (one unit of alcohol equals 250 ml beer, 125 ml wine or 25 ml spirits) or recovered alcoholics
* Regular consumption of beverages or food containing methylxanthines (e.g. coffee, tea, cola, caffeine containing sodas, chocolate) equivalent to more than 500 mg methylxanthines per day
* Positive drug screening and/or positive alcohol test at entry screening or on hospitalization day -1
* Pregnant and/or nursing women. Positive pregnancy test at entry screening or on hospitalization day -1
* Allergic diathesis or any clinically significant allergic disease (i.e. asthma or bronchial hyperreactivity)
* Known allergy to sticking plaster or to the ingredients of the products
* History of or active skin disease or dermatologic disease that might interfere with the evaluation of test site reaction
* Any history of drug hypersensitivity (especially to the active and inactive ingredients of the ibuprofen preparations and NSAIDs including subjects where attacks of asthma, angioedema, urticaria or rhinitis have been precipitated), or intolerance to any sugar (e.g. fructose, glucose, or lactose)
* History of clinically significant food allergies or current significant or perennial allergy at screening
* History of autoimmune disorders such as lupus erythematosus
* Presence or a history of clinically significant cardiovascular, renal, hepatic, pulmonary, metabolic, endocrine, haematological, gastrointestinal, neurological, psychiatric or other diseases
* Clinically significant illness within 4 weeks before entry screening and during the study
* Major surgery of the gastrointestinal tract except for appendectomy
* Any chronic disease which might interfere with absorption, distribution, metabolism or excretion of the drug
* Intensive UV-light exposure (sunbaths) at the application site or use of tanning beds within 2 weeks before entry screening and during the study
* Intake or administration of any systemic or any topical medication (including immune system interfering drugs, OTC medication and especially intake of antacids e.g. aluminum hydroxide, magnesium hydroxide, and simethicone or herbal medication e.g. St. John's wort, kava kava, or use of ointments, gels or patches for skin application, piperine containing products16) as well as hormone replacement therapy within 2 weeks before entry screening and during the study, except single doses of paracetamol given in case of an adverse event (e.g. headache) during the study
* Use of topical products without medication at the application sites (including make-up, sunscreen, creams, lotions, powders, alcohol) 7 days prior to entry screening until discharge
* Administration of depot injectable solutions or medications with a half-life > 1 week (including study medications) within 6 months before entry screening
* Intake of enzyme-inducing, organotoxic or long half-life drugs within 4 weeks before entry screening
* Medication with drugs known to alter the major organs or systems such as barbiturates, phenothiazines, cimetidine, omeprazole etc. within the last 2 months prior entry screening
* Any method of hair removal (e.g. waxing, shaving, epilating, laser) at the application sites 7 days prior to entry screening until discharge
* Subjects with tattoos, sunburn, coloration, open sores or scars (e.g. any burning or stinging) on site(s) of application
* History of difficulty in swallowing
* Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies
* Systolic blood pressure outside the range of 100 to 140 mmHg and/or diastolic blood pressure outside the range of 60 to 90 mmHg17 at entry screening visit
* Heart rate outside the range of 50 to 90 beats/min at entry screening visit
* Respiratory rate outside the range of 12-24 breaths/min at entry screening visit
* Axillary body temperature outside the interval of 35.5 to 37.1°C at entry screening visit
* Any clinically significant abnormality of the resting ECG (12-lead) (i.e. AV block, 2° to 3°, sinus bradycardia, sick sinus syndrome, SA block)
* Laboratory values outside normal range with clinical relevance at entry screening visit
* Vomiting within the first 4 hours after dosing with oral ibuprofen
* Diarrhoea within the first 24 hours after dosing with oral ibuprofen
* Special diet due to any reason, e.g. vegetarians
* Not fulfilling study specific restrictions given in a study protocol
* Engagement in strenuous exercise within 2 weeks prior to check-in (e.g., marathon runners, weight lifters)
* Subjects who are known or suspected:
* not to comply with the study directives
* not to be reliable or trustworthy
* not to be capable of understanding and evaluating the information given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed
* to be in such a precarious financial situation that they no longer weigh up the possible risks of their participation and the inconvenience they may be involved in
* subject is a dependent person, e.g. a relative, family member, or member of the investigator's or sponsor's staff
* subject is in custody or submitted to an institution due to a judicial order.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
AUC(0-12h) of ibuprofen | 5 days
  Area under the concentration/time curve, from time 0 h to 12 h
AUC(0-t) of Ibuprofen | 5 days
  Area under the concentration/time curve, calculated by the trapezoidal rule from time 0 h to last observed concentration at time t
Cmax of Ibuprofen | 5 days
  Observed maximal concentration after administration

SECONDARY OUTCOMES:
Tmax after multiple dosing | 5 days
  Observed time point of maximal concentration
t½ after multiple dosing | 5days
  Plasma concentration half-life calculated according to t1/2=ln(2)/ λz
λz of total ibuprofen after multiple dosing | 5 days
  Terminal rate constant (slowest rate constant of the disposition) negative of the slope of a log-linear regression of the unweighted data considering the last concentration-time points ≥ LLOQ
AUC(0-inf) after multiple dosing | 5 days
  Area under the concentration/time curve, from time 0 h extrapolated to infinity (AUC(0-∞) = AUC(0-t) + Clast/λz where Clast is the last concentration above the limit of quantification and λz is the terminal elimination constant)

OTHER OUTCOMES:
AUC(0-τ) After plaster removal, | 5 days
  Area under the concentration/time curve, from time 0 h the end of the treatment period
Number of subjects with product related Adverse Events | 15 days
  Adverse events from subject informed consent until the follow-up call
Change in dermal effect score to baseline | 15 days
  Skin irritation by using "Dermal Effect Score" and "Other Effect Score") Dermal Response Score Score Definition 0- No evidence of irritation
  1. - Minimal erythema, barely perceptible
  2. - Definite erythema, readily visible; minimal oedema or minimal papular
  3. - Erythema and papules
  4. - Definite oedema
  5. - Erythema, oedema, and papules
  6. - Vesicular eruption
  7. - Strong reaction spreading beyond test site
  Score Definition 0 - None observed
  1. - Slight glazed appearance
  2. - Marked glazing
  3. - Glazing with peeling and cracking
  4. - Glazing with fissures. Film of dried serous exudates covering all or part of the patch site Small petechial erosions and/or scabs
Abnormal laboratory findings | 15 days
  Abnormal laboratory findings with respect to the pre-defined reference ranges
Adhesion (quantitative, using the mean adhesion score) and qualitative assessment of the plaster | Day 1 and Day 5
  The percentage of the Ibuprofen 200 mg TEPI plaster adhered to the skin will be assessed at the following time points on application of plaster 1 and plaster 5: at placement of plaster (T0) and then at the following time points post placement: 4, 8, 12, 16, 20 and 24 hours. An adhesion score will be assigned using a 5-point numerical scale 0 = ≥ 90% adhered (essentially no lifting off the skin)
  1. = ≥ 75% to < 90% adhered (some edges only lifting off the skin)
  2. = ≥ 50% to < 75% adhered (less than half of the plaster lifting off the skin)
  3. = > 0% to < 50% adhered (not detached, but more than half of the plaster lifting off the skin without falling off)
  4. = 0% adhered (plaster detached; completely off skin)
Cmax, ss after plaster removal | 5 days
  Observed maximal concentration after administration at steady state
CT, ss after plaster removal | 5 days
  Observed maximal concentration after administration at the end of τ at steady state
residual ibuprofen in removed plasters | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of Clinical Pharmacology and Therapeutics University Multidisciplinary Hospital for Active Treatment 'Tsaritsa Ioanna-ISUL' EAD, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No